CLINICAL TRIAL: NCT01994083
Title: A Double-blind, Randomised, Placebo-controlled, Parallel Group, Dose Escalation Study to Investigate the Safety, Tolerability and Pharmacokinetics of Multiple Oral Doses of IX-01 in Healthy Male Subjects
Brief Title: A Study of Multiple Oral Doses of IX-01 in Healthy Men
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ixchelsis Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IX-0101
Record Dates: First submitted 2013-11-19; First posted 2013-11-25 (Estimated); Last update posted 2014-09-03 (Estimated); Status verified 2014-09

CONDITIONS: Healthy Participants

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo
- IX-01 (Experimental): Up to 4 different dose groups within 50 to 1,200 mg of IX-01 oral aqueous dispersion, administered once daily for 10 days
  Interventions: Drug: IX-01

INTERVENTIONS:
Drug: Placebo — Administered orally
  Arms: Placebo
Drug: IX-01 — Administered orally
  Arms: IX-01

SUMMARY:
The purpose of this study is to investigate the safety and tolerability of IX-01 after multiple doses, and to determine how the body handles IX-01.

ELIGIBILITY:
Inclusion Criteria:

* A body mass index (Quetelet index) in the range 18-30
* Total body weight greater than (>)50 kilograms (kg) at screening
* Able to understand the nature of the trial and any hazards of participating in it
* Able to communicate satisfactorily with the investigator and to participate in, and comply with the requirements of, the entire trial
* Participants and their partners must be willing to use adequate forms of contraception and comply with contraception requirements during the trial, and for 4 months after the last dose of medication
* Must not plan to donate sperm or father a child during the trial, and for 4 months after the final dose of medication

Exclusion Criteria:

* Clinically relevant abnormal history, physical findings, electrocardiogram (ECG), or laboratory values at the screening assessment that could interfere with the objectives of the trial or the safety of the participant
* Presence of acute or chronic illness or history of chronic illness sufficient to invalidate participation in the trial or make it unnecessarily hazardous
* Impaired gastrointestinal, endocrine, thyroid, hepatic, cardiovascular, respiratory, haematological, renal or neurological function, diabetes mellitus, coronary heart disease, or history of any psychotic mental illness
* Surgery (for example (e.g.) stomach bypass) or medical condition that might affect absorption, metabolism or elimination of medicines
* Presence or history of severe adverse reaction to any drug
* Use of any prescription or over-the-counter medicine during the 14 days before the first dose of trial medication, or intention to use any medicine during the trial, with the exception of short courses of medication considered by the investigator not to interfere with the safety of the participant or the integrity of the trial data (such as acetaminophen (paracetamol))
* Current use of any herbal remedy or nutritional supplement, or intention to use any such product during the study
* Participation in another clinical trial of a new chemical entity or a prescription medicine within the previous 3 months
* Previous participation in this trial or any other clinical trial of an oxytocin receptor antagonist
* Presence or history of drug or alcohol abuse, or intake of more than 21 units of alcohol weekly or more than 5 cigarettes daily
* Blood pressure and heart rate in supine position at the screening examination outside the ranges 90-130 millimeters of mercury (mm Hg) systolic, 50-90 mm Hg diastolic; heart rate 50-90 beats/minute
* Possibility that the participant will not cooperate with the requirements of the protocol
* Evidence of drug abuse on urine testing
* Positive test for hepatitis B, hepatitis C, Human Immunodeficiency Virus 1(HIV1) or Human Immunodeficiency Virus 2 (HIV2)
* Loss of more than 400 milliliters (mL) blood during the 3 months before the trial, e.g. as a blood donor
* Objection by General Practitioner (GP), on medical grounds, to participant entering trial

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2013-11; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Number of Participants with One or More Drug Related Adverse Events (AEs) or any Serious AEs | Baseline to Day 20 (Estimated up to 3 weeks)

SECONDARY OUTCOMES:
Peak Plasma Concentration (Cmax) of IX-01 | Pre-dose to 24 hours post dose on Days 1 and 10
Area Under the Plasma Concentration-Time Curve (AUCtau) | Pre-dose up to 24 hours post dose on Days 1 and 10
Time of Peak Plasma Concentration (Tmax) of IX-01 | Pre-dose to 24 hours post dose on Days 1 and 10
Elimination Half Life (t1/2) of IX-01 | Pre-dose up to 96 hours post dose on Day 10
Accumulation Ratio (Racc) of IX-01 based on AUCtau | Pre-dose up to 24 hours post dose on Day 10
Accumulation Ratio (Racc) of IX-01 based on Cmax | Pre-dose up to 24 hours post dose on Days 1 and 10
Area Under the Concentration-Time Curve (AUCt) from Zero to the Time of Last Quantifiable Concentration (AUC(0-t)) of IX-01 | Pre-dose to 96 hours post dose on Day 10
Minimum Observed Concentration (Ctrough) of IX-01 | Pre-dose on Days 2 to 10
Elimination Rate Constant (Kel) of IX-01 | Pre-dose up to 96 hours post dose on Day 10
Apparent Clearance of IX-01 | Pre-dose up to 24 hours post dose on Day 10
Apparent Volume of Distribution During the Terminal Phase of IX-01 | Pre-dose up to 96 hours post dose on Day 10
Urine 6-β-hydroxycortisol/cortisol Ratio | Pre-dose on Day 1 and Day 10
IX-01 Concentration and Amount Secreted in Semen | Between 2 and 4 hours after dosing, on Day 9

CONTACTS AND LOCATIONS:
Overall Officials: Email: Ixchelsis@Choruspharma.com, Study Director — Ixchelsis Limited
Locations (1):
- Hammersmith Medicines Research (HMR), London, United Kingdom